CLINICAL TRIAL: NCT02719106
Title: Evaluation of Effectiveness and Safety of Ultimaster® Stent in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: IRIS Ultimaster Cohort in the IRIS-DES Registry
Acronym: IRISUltimaster
Status: Completed | Type: Observational
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Sponsor-investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2016-05
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: real world data; percutaneous coronary intervention; drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultimaster stent
  Interventions: Device: Ultimaster stent

INTERVENTIONS:
Device: Ultimaster stent

SUMMARY:
The purpose of this study is to evaluate the relative effectiveness and safety of Ultimaster stent compared to other drug eluting stents.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Intervention with Ultimaster stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with Ultimaster stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Ultimaster stent
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Composite event | 1year
  The number of events with the first occurrence of a composite event(death, non-fatal myocardial infarction, target vessel revascularization)

SECONDARY OUTCOMES:
All death | 5years
Cardiac death | 5years
Myocardial infarction | 5years
Composite event of death or myocardial infarction | 5years
Composite event of cardiac death or myocardial infarction | 5years
Target Vessel revascularization | 5years
  Defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself. Clinical-driven Clinically indicated angiography at follow-up shows a percent diameter stenosis ≥ 50% (core lab QCA assessment) and if one of the following occurs: (1) a positive history of recurrent angina pectoris, presumably related to the target vessel; (2) objective signs of ischemia at rest (ECG changes) of during exercise test (or equivalent), presumably related to the target vessel; (3) abnormal results of any invasive functional diagnostic test (eg, Doppler flow velocity reserve, fractional flow reserve). Ischemia-driven if one of followings of above-mentioned symptom (clinical-driven) or sign of ischemia or diameter stenosis ≥ 70 %
Target Lesion revascularization | 5years
  Defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLRs should be classified prospectively as clinically indicated or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Stent thrombosis | 5years
  DEFINITE stent thrombosis : acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE stent thrombosis : unexplained death within 30 days or target-vessel infarction without angiographic information Academic Research Consortium (ARC) stent thrombosis is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute stent thrombosis: 0-24 hours after stent implantation; Subacute stent thrombosis: >24 hours to 30 days post; late stent thrombosis: >30 days to 1 year post; Very late stent thrombosis: >1 year post;
Stroke | 5years
Procedural success | 3days
  Defined as mean lesion diameter stenosis ≤50% and without the occurrence of in-hospital myocardial infarction (MI), target vessel revascularization (TVR), or death

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Sejong General hospital, Bucheon-si
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Gangneung Asan Hospital, Gangneung
  - Inje University Ilsan Paik Hospital, Ilsan
  - Kwangju Christian Hospital, Kwangju
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's hospital, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided